CLINICAL TRIAL: NCT05308498
Title: Retrospective Evaluation to Compare Small Bowel Video Reading by AKE-1 (Navicam SB) Capsule Endoscope System With and Without ProScan Module and PillCam SB3 Capsule System With SBI
Brief Title: Retrospective Evaluation to Compare AKE-1 (Navicam SB) Capsule Endoscope System and PillCam SB3 Capsule System
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 102-CEP-0002
Record Dates: First submitted 2022-03-06; First posted 2022-04-04 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Retrospective Study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESView software with ProScan: evaluate the performance of the NaviCam SB Capsule System ProScan software feature in comparison with the PillCam SB3 Capsule system SBI feature
  Interventions: Diagnostic Test: ESView software with proscan
- Rapid software with SBI: evaluate the performance of the NaviCam SB Capsule System ProScan software feature in comparison with the PillCam SB3 Capsule system SBI feature
  Interventions: Diagnostic Test: Rapid software with SBI

INTERVENTIONS:
Diagnostic Test: ESView software with proscan — Each reviewer will review random video and record all lesions/findings with the ESView software with ProScan.
  Groups: ESView software with ProScan
Diagnostic Test: Rapid software with SBI — Each reviewer will review random video and record all lesions/findings with the PillCam Rapid software with SBI.
  Groups: Rapid software with SBI

SUMMARY:
This is a retrospective study on prospectively collected patient video data from a multicenter, single-blinded pivotal trial (Ethics Approval No. [2021] (0635-01)), involving a consecutive series of patients recruited by 3 Chinese centers based on the suspected small bowel disease, gastrointestinal bleeding, etc. All video images will be anonymized (de-identified). Video images from both the investigational device and comparator device are reviewed by two independent reviewers. Once the conventional reading has been completed, each reviewer will then review randomized videos with the ProScan feature enabled in ESView or SBI enabled on the Pillcam Rapid software. Each reviewer should review for normal versus abnormal findings, type of visual findings and categorization (lesions, polyps, bleeding, etc.), diagnosis, reading time, and subjective assessment of visual quality.

DETAILED DESCRIPTION:
This is a retrospective study on prospectively collected patient video data from a multicenter, single-blinded pivotal trial, involving a consecutive series of patients recruited by 3 Chinese centers based on the suspected small bowel disease, gastrointestinal bleeding, etc.

Video images from both the investigational device and comparator device are reviewed by two independent reviewers. Video that will be retrospectively collected, have been anonymized. Each reviewer will review the images collected according to the "conventional reading" as recommended by ACG guidelines.

Once the conventional reading has been completed, each reviewer will then review randomized videos with the ProScan feature enabled in ESView or SBI enabled on the Pillcam software . Each reviewer will then review the videos and document all lesions/findings found by the ProScan and Pillcam software with SBI. Annotations should be done after the reading, each finding shall be labelled and categorized (active bleeding, Angioectasia, polyps/ nodules, tumors or varisces, ulcers, isolated erosions, lesions, other).

For all lesions/findings, if there was significant disagreement between two reviewers for the same image, for both capsule videos, another independent reviewer will then review the video of that examination and provide his review results.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in the study titled Performance Evaluation of the NaviCam SB Capsule Endoscope System in Comparison to the PillCam SB3 Capsule System for the Diagnosis of Small Bowel Diseases (Ethics Approval No. [2021] (0635-01)) and were included in the FAS.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who participated in the study titled Performance Evaluation of the NaviCam SB Capsule Endoscope System in Comparison to the PillCam SB3 Capsule System for the Diagnosis of Small Bowel Diseases (Ethics Approval No. [2021] (0635-01)) and were included in the FAS.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic consistency | 1 month
  The agreement rate between ESView software with ProScan assisted reading mode in the AKE-1 system and Rapid software with SBI pre-selection mode in the PillCam SB3 system on video classification, i.e. normal or abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: XiaoHua Hou, Principal Investigator — Union Hospital of Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Union Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No